CLINICAL TRIAL: NCT03095612
Title: An Investigator-sponsored, Phase 1/2 Trial of the Oral XPO1 Inhibitor Selinexor (KPT-330) Monotherapy and in Combination With Docetaxel for Previously Treated, Advanced KRAS Mutant Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase 1/2 Trial of Selinexor (KPT-330) With Docetaxel for Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding Sponsor no longer supporting study
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, David E Gerber, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 032017-003
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — selinexor; Docetaxel

STUDY DESIGN:
Intervention Model Description: Docetaxel will be given once every 3 weeks. Treatment will be administered in 21-day cycles. Dose limiting toxicities (DLTs) will be assessed based on the first cycle (7-day lead-in plus 21-day cycle = 28 days) toxicity using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03. A standard 3 + 3 dose escalation paradigm will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor Monotherapy and in Combination with Docetaxel (Experimental): For the selinexor monotherapy cohort, 6 patients each will be treated in two dosing cohorts (weekly and biweekly). Selinexor once weekly oral (40mg, 60mg, 80mg) OR Selinexor twice weekly oral (60mg, 40mg, 60mg weekly).
  Selinexor will be administered once weekly starting one week before chemotherapy initiation in combination with docetaxel. Docetaxel will be given once every 3 weeks. Treatment will be administered in 21-day cycles. Selinexor dose escalation: 60, 80, 40 mg once weekly. Docetaxel 75 mg/m2 IV, 60 every 3 weeks.
  Interventions: Drug: Selinexor; Drug: Docetaxel

INTERVENTIONS:
Drug: Selinexor — Selinexor once weekly oral or twice weekly oral
  Other Names: KPT-330
Drug: Docetaxel — Docetaxel once every 3 weeks (75 mg/m2 IV)

SUMMARY:
This study is being done to evaluate the safety of the investigational study drug, selinexor when given with docetaxel to patients who have been previously treated for advanced KRAS mutant lung cancer.

DETAILED DESCRIPTION:
This is a phase 1/2 single-arm, non-blinded, multi-institutional study. Selinexor will be administered once weekly starting one week before chemotherapy initiation (to permit pharmacodynamic assessment of selinexor alone and in combination with chemotherapy).This study will compare safety and outcomes with historical controls (docetaxel monotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

  1. Written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure. However, the Investigator should not repeat procedures that are performed as part of standard of care (SOC), if they are within the screening window and are done prior to signing the ICF.
  2. Age ≥ 18 years
  3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
  4. Histologically or cytologically confirmed advanced (stage 4, according to the American Joint Committee on Cancer [AJCC] version 7.0 Staging manual) NSCLC
  5. Molecular identification of a KRAS mutation (codons 12, 13, or 61 mutations detected by sequencing) by a CLIA-certified assay (source documentation required).
  6. Tissue available for analysis at time of enrollment for biomarker analysis: 10 unstained slides plus 1 H+E slide. If archival tumor tissue is not available in select cases, subjects may be permitted to enroll on the study with prior approval of the study PI.
  7. At least one and up to two previous lines of systemic cytotoxic therapy for advanced NSCLC, of which one must have been a platinum-based doublet therapy. Up to four total previous lines of systemic therapy (including immunotherapy and molecularly targeted therapy) for advanced NSCLC.
  8. Radiographic or clinical disease recurrence or progression during or after the last line of systemic therapy
  9. Adequate hematologic function (absolute neutrophil count [ANC] ≥ 1500 cells/µL; hemoglobin ≥ 9 g/dL; platelets ≥ 100,000/µL. Patients may be transfused with PRBCs up to 7 days prior to when enrollment labs are drawn to achieve Hgb ≥9.0 mg/dL.
  10. Adequate renal function (calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation)
  11. Adequate hepatic function (total bilirubin ≤ upper limit of normal [ULN], alanine aminotransferase [ALT] ≤ 2 × ULN and aspartate aminotransferase [AST] ≤ 2 × ULN). ALT and/or AST may be ≤ 5 × ULN if due to liver metastases. If ALT or AST is > 2 and ≤ 5 × ULN in patients with liver metastases, alkaline phosphatase must be ≤ 2.5 × ULN (unless elevated alkaline phosphatase clearly due to skeletal-rather than hepatic-process; eg, normal GGT, presence of multiple bone metastases, absence of bulky and/or central liver metastases). Patients with Gilbert's syndrome are allowed if total bilirubin ≤ 2 × ULN and direct bilirubin is ≤ ULN.
  12. Female patients of childbearing potential must agree to use 2 methods of contraception (including 1 highly effective and 1 effective method of contraception) and have a negative serum pregnancy test at Screening. Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose of study treatment. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use 2 reliable methods of contraception throughout the study and for 3 months after their last dose of medication. Female patients are considered NOT of childbearing potential if they have a history of surgical sterility (including hysterectomy and/or bilateral oophorectomy, but not tubal ligation alone) or evidence of post-menopausal status defined as any of the following:

      * Natural menopause with last menses >1 year ago
      * Radiation-induced oophorectomy with last menses >1 year ago
      * Chemotherapy-induced menopause with last menses >1 year ago.

      Male patients and their partners must use 2 reliable methods of contraception, at least one of them a barrier method (if sexually active with a female of child-bearing potential).
  13. Measurable disease according to RECIST v1.1
  14. Previously treated (surgery and/or radiation therapy) or untreated brain metastases are eligible, provided that patients are asymptomatic and not requiring escalating doses of corticosteroids.
  15. Previous treatment-associated clinically significant toxicities resolved to CTCAE grade ≤2 (except alopecia) or to their baseline. NOTE: Prior immunotherapy-related endocrinopathy controlled with ongoing medical management (eg, hypothyroidism, adrenal insufficiency, diabetes) is permitted
  16. At least 3 weeks or 5 half-lives, whichever is shorter, since receiving systemic anticancer therapy, including investigational agents, prior to starting study therapy. At least 2 weeks since receiving radiation therapy prior to starting study therapy

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

  1. Patients who are pregnant or lactating
  2. Major surgery (excluding skin biopsies and procedures for insertion of central venous access devices) within 2 weeks of first dose of study drug
  3. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety
  4. Concurrent active malignancy that would interfere with treatment administration or assessment in the opinion of the treating investigator
  5. Unstable cardiovascular function:

     * Symptomatic ischemia, or
     * Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmics is excluded; 1st degree AV block or asymptomatic LAFB/RBBB are not excluded; asymptomatic rate controlled atrial fibrillation is not excluded), or
     * Congestive heart failure (CHF) of NYHA Class ≥3, or
     * Myocardial infarction (MI) within 3 months
  6. Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; however, prophylactic use of these agents is acceptable even if parenteral
  7. Pre-existing grade 3 or 4 neuropathy
  8. Active Hepatitis A, B or C infection
  9. Known human immunodeficiency virus (HIV) infection (HIV testing is not required as part of this study)
  10. Patients unable to swallow tablets, patients with malabsorption syndrome, or any other GI disease or GI dysfunction that could interfere with absorption of study treatment
  11. Prior exposure to docetaxel, selinexor, or another selective inhibitor of nuclear transport (SINE) compound (NOTE: prior docetaxel exposure permitted in selinexor monotherapy cohort)
  12. Patients unwilling to comply with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Pittsburgh Medical Center-Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Vanderbilt Medical Center-Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 subjects consented;1 screen failed prior to receiving treatment. Participants started at dosing selinexor 60 mg + docetaxel 75 mg/m2. The second dose level was 80 mg +docetaxel 75 mg/m2 to which 4 subjects were assigned. Then 33 patients enrolled and started on Dose expansion: selinexor 60 mg weekly plus docetaxel 75 mg/m2 3 weekly. No data was collected or analyzed for the selinexor Monotherapy cohort, study was halted due to funding.
Groups:
- Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel; Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel; Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel: '3x3' Dose escalation (cycle = 21 days). Selinexor once weekly oral administration (cohorts 60mg, 80mg, 100mg…) Docetaxel once every 3 weeks (75mg/m2 IV).
  cohort escalation until MTD (maximum tolerated dose) is established.
- Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel: Selinexor once weekly oral administration Docetaxel once every 3 weeks (75 mg/m2 IV)
- Selinexor 40 mg Monotherapy; Selinexor 60 mg Monotherapy; Selinexor 80 mg Monotherapy: Selinexor once weekly oral (40mg, 60mg, 80mg)
  OR
  Selinexor twice weekly oral (40mg, 60mg, 80mg)
Period: Dose Escalation:Selinexor 60mg+Docetaxel
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Escalation:Selinexor 80mg+Docetaxel
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 0 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Dose not tolerated by the subject | 0 | 4 | 0 | 0 | 0 | 0 | 0
Period: Dose Escalation:Selinexor100mg+Docetaxel
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion:Selinexor 60 mg+Docetaxel
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 0 | 0 | 0 | 33 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 33 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Selinexor 40 mg Monotherapy
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Selinexor 60 mg Monotherapy
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Selinexor 80 mg Monotherapy
Arm/Group | Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 80 mg and in Combination With Docetaxel | Dose Escalation Phase: Selinexor 100 mg and in Combination With Docetaxel | Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 41 subjects were consented, but 1 screen failed and only 40 total were assigned to combination treatment cohort. 2nd dose level of 80 mg +docetaxel 75 mg/m2 was not tolerated and hence did not proceed to next dose of 100 mg+ docetaxel 75 mg/m2 as well. The study was halted prior to participants receiving any of the selinexor monotherapy. No data was collected or analyzed for the selinexor Monotherapy cohort.
Groups:
- Dose Escalation: Selinexor 60 mg + Docetaxel: Dose Escalation Phase: Selinexor 60 mg and in Combination With Docetaxel '3x3' Dose escalation (cycle = 21 days). Selinexor once weekly oral administration (cohorts 60mg, 80mg) Docetaxel once every 3 weeks (75mg/m2 IV).
  cohort escalation until MTD (maximum tolerated dose) is established.
- Dose Escalation: Selinexor 80 mg + Docetaxel: Dose Escalation Phase: Selinexor 800 mg and in Combination With Docetaxel '3x3' Dose escalation (cycle = 21 days). Selinexor once weekly oral administration (cohorts 60mg, 80mg) Docetaxel once every 3 weeks (75mg/m2 IV).
  cohort escalation until MTD (maximum tolerated dose) is established.
- Dose Expansion Phase: Selinexor 60 + Docetaxel: Dose Expansion Phase: Selinexor 60 mg and in Combination With Docetaxel Selinexor once weekly oral administration Docetaxel once every 3 weeks (75 mg/m2 IV)
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Selinexor 60 mg + Docetaxel | Dose Escalation: Selinexor 80 mg + Docetaxel | Dose Expansion Phase: Selinexor 60 + Docetaxel | Total
Number analyzed (Participants) | 3 | 4 | 33 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 18 | 20
  >=65 years | 2 | 3 | 15 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 17 | 23
  Male | 0 | 1 | 16 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 32 | 39
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 1 | 4
  White | 0 | 3 | 30 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 33 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: A DLT was any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0). DLTs were collected to determine the Maximum-Tolerated Dose (MTD).
  **DLT will include the following when considered to be at least possibly related to study drug administration: 1) > 1 missed doses (out of 4 doses) of study treatment during cycle 1 due to study treatment related toxicities 2) Discontinuation of study therapy before completion of Cycle 1, due to study-drug related toxicity.
Time Frame: Each 21 day cycle for 2 years
Population: The study was halted prior to participants receiving selinexor monotherapy. No data was collected or analyzed for the selinexor Monotherapy Cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Selinexor in Combination With Docetaxel Cohort: Selinexor will be administered once weekly starting one week before chemotherapy initiation in combination with docetaxel. Docetaxel will be given once every 3 weeks. Treatment will be administered in 21-day cycles. Selinexor dose escalation: 60, 80, 40 mg once weekly. Docetaxel 75 mg/m2 IV, 60 every 3 weeks.
  Selinexor: Selinexor once weekly oral or twice weekly oral
  Docetaxel: Docetaxel once every 3 weeks (75 mg/m2 IV)
- Selinexor Monotherapy Cohort: For the selinexor monotherapy cohort, 6 patients each will be treated in two dosing cohorts (weekly and biweekly). Selinexor once weekly oral (40mg, 60mg, 80mg) OR Selinexor twice weekly oral (60mg, 40mg, 60mg weekly).
Arm/Group | Selinexor in Combination With Docetaxel Cohort | Selinexor Monotherapy Cohort
Number analyzed (Participants) | 40 | 0
Participants
  selinexor, 80 mg | 3 | 0
  selinexor, 60 mg | 37 | 0

2. Secondary Outcome: Tumor Size Will be Assessed Using the RECIST v1.1
Description: To evaluate the efficacy of selinexor monotherapy and in combination with docetaxel in patients with advanced KRAS mutant NSCLC. Tumor size will be assessed at baseline and every 2 cycles (ie, after 7 weeks for first 2 cycles, and then every 6 weeks) during the treatment period using the Response Evaluation Criteria in Solid Tumors RECIST v1.1 criterion.
Time Frame: Each 21 day cycle for 2 years
Population: 32 patients were evaluable for disease. This was a 3+3 dose escalation study, participants started at dosing selinexor 60 mg + docetaxel 75 mg/m2. Dose tolerated for 3 patients. 2nd dose level of 80 mg +docetaxel 75 mg/m2 was not tolerated and data was not collected. The remainder of the patients enrolled were then started on selinexor 60 mg weekly plus docetaxel 75 mg/m2 3 weekly. No data was collected or analyzed for the selinexor Monotherapy cohort, study was halted due to funding.
Measure: Count of Participants; unit: Participants
Groups:
- Selinexor 60 mg and in Combination With Docetaxel; Selinexor 80 mg and in Combination With Docetaxel; Selinexor 100 mg and in Combination With Docetaxel: '3x3' Dose escalation (cycle = 21 days). Selinexor once weekly oral administration (cohorts 60mg, 80mg, 100mg…) Docetaxel once every 3 weeks (75mg/m2 IV).
  cohort escalation until MTD (maximum tolerated dose) is established.
Arm/Group | Selinexor 60 mg and in Combination With Docetaxel | Selinexor 80 mg and in Combination With Docetaxel | Selinexor 100 mg and in Combination With Docetaxel | Selinexor 40 mg Monotherapy | Selinexor 60 mg Monotherapy | Selinexor 80 mg Monotherapy
Number analyzed (Participants) | 32 | 0 | 0 | 0 | 0 | 0
Participants | 25 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of time over 4 years, 7 months.
Description: No data collected or analyzed for monotherapy as the study was halted early due to funding.
Groups:
- Dose Escalation: Selinexor 60mg + Docetaxel 75mg/m2; Dose Escalation: Selinexor 80mg + Docetaxel 75mg/m2; Dose Escalation:Selinexor 100mg + Docetaxel 75mg/m2: Selinexor will be administered once weekly starting one week before chemotherapy initiation in combination with docetaxel. Docetaxel will be given once every 3 weeks. Treatment will be administered in 21-day cycles. Selinexor dose escalation: 60, 80, 100 mg once weekly. Docetaxel 75 mg/m2 IV, 60 every 3 weeks.
  Selinexor: Selinexor once weekly oral or twice weekly oral
  Docetaxel: Docetaxel once every 3 weeks (75 mg/m2 IV)
- Dose Expansion: Selinexor 60 mg + Docetaxel 75mg/m2: Selinexor dose escalation: 60mg once weekly. Docetaxel 75 mg/m2 IV, 60 every 3 weeks.
- Selinexor 40mg Monotherapy; Selinexor 60mg Monotherapy; Selinexor 80mg Monotherapy: For the selinexor monotherapy cohort, 6 patients each will be treated in two dosing cohorts (weekly and biweekly). Selinexor once weekly oral (40mg, 60mg, 80mg) OR Selinexor twice weekly oral (60mg, 40mg, 60mg weekly).
Arm/Group | Dose Escalation: Selinexor 60mg + Docetaxel 75mg/m2 | Dose Escalation: Selinexor 80mg + Docetaxel 75mg/m2 | Dose Escalation:Selinexor 100mg + Docetaxel 75mg/m2 | Dose Expansion: Selinexor 60 mg + Docetaxel 75mg/m2 | Selinexor 40mg Monotherapy | Selinexor 60mg Monotherapy | Selinexor 80mg Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/0 | 0/33 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/4 | 0/0 | 0/33 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 0/0 | 33/33 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Selinexor 60mg + Docetaxel 75mg/m2 (N=3) | Dose Escalation: Selinexor 80mg + Docetaxel 75mg/m2 (N=4) | Dose Escalation:Selinexor 100mg + Docetaxel 75mg/m2 (N=0) | Dose Expansion: Selinexor 60 mg + Docetaxel 75mg/m2 (N=33) | Selinexor 40mg Monotherapy (N=0) | Selinexor 60mg Monotherapy (N=0) | Selinexor 80mg Monotherapy (N=0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Laceration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets Decreased (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypoxia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Selinexor 60mg + Docetaxel 75mg/m2 (N=3) | Dose Escalation: Selinexor 80mg + Docetaxel 75mg/m2 (N=4) | Dose Escalation:Selinexor 100mg + Docetaxel 75mg/m2 (N=0) | Dose Expansion: Selinexor 60 mg + Docetaxel 75mg/m2 (N=33) | Selinexor 40mg Monotherapy (N=0) | Selinexor 60mg Monotherapy (N=0) | Selinexor 80mg Monotherapy (N=0)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (8) | 1 (1) | 0 (0) | 21 (44) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (6) | 2 (8) | 0 (0) | 23 (47) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 19 (24) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (9) | 1 (1) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 0 (0) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (9) | 3 (11) | 0 (0) | 11 (20) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Lymphocytes Decreased/Lymphopenia/Leukopenia (Investigations) | 3 (16) | 3 (11) | 0 (0) | 7 (16) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (6) | 0 (0) | 8 (16) | 0 (0) | 0 (0) | 0 (0)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (12) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Platelet Counts Decreased (Investigations) | 1 (2) | 1 (3) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (4) | 1 (1) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 4 (16) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (15) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (13) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (14) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (7) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT03095612/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03095612/ICF_001.pdf